CLINICAL TRIAL: NCT01091597
Title: PV Isolation Versus Box Isolation for the Treatment of Atrial Fibrillation
Brief Title: Pulmonary Vein (PV) Isolation Versus Box Isolation for the Treatment of Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Charles Henrikson, MD, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00008424
Record Dates: First submitted 2010-03-23; First posted 2010-03-24 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2010-03

CONDITIONS: Atrial Fibrillation; Radiofrequency Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- usual ablation (Active Comparator): Wide-area circumferential ablation of the pulmonary veins
  Interventions: Procedure: usual PV ablation
- Box isolation of the pulmonary veins (Experimental): Single Box lesion set encompassing all four pulmonary veins and the posterior wall of the left atrium.
  Interventions: Procedure: Box isolation of pulmonary veins

INTERVENTIONS:
Procedure: usual PV ablation — usual PV ablation, per above
  Arms: usual ablation
Procedure: Box isolation of pulmonary veins — as above
  Arms: Box isolation of the pulmonary veins

SUMMARY:
Curative catheter ablation has been established as an effective therapeutic option for atrial fibrillation (AF) that is resistant to pharmacologic rhythm or rate control. However, standard ablative approaches targeting the pulmonary veins (PVs) are associated with a success rate as low as 40%. In a recent study, Kumagai et al. described a new approach of catheter ablation of AF isolating the posterior left atrium including all PVs (called Box Isolation). In Kumagai's study, 46 patients with symptomatic AF underwent box isolation. At 6 months follow up, 43 of 46 patients (93%) were arrhythmia free without antiarrhythmic drugs, with a single procedure success rate of 87% (40/46). This study provided new evidence supporting the hypothesis that the posterior wall is of high importance for the maintenance of AF. The aim of the investigators study is to determine the efficacy of two different approaches of catheter ablation (Standard PV Isolation vs. Box isolation) for the treatment of chronic AF.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing clinically indicated pulmonary vein ablation for atrial fibrillation.

Exclusion Criteria:

* Unable to understand consent form. Not scheduled for clinically indicated pulmonary vein ablation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-06; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
freedom from atrial fibrillation | 3 months following ablation

SECONDARY OUTCOMES:
safety of Box isolation | 3 months following procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Chilukuri K, Scherr D, Dalal D, Cheng A, Spragg D, Nazarian S, Barcelon BD, Marine JE, Calkins H, Henrikson CA. Conventional pulmonary vein isolation compared with the "box isolation" method: a randomized clinical trial. J Interv Card Electrophysiol. 2011 Nov;32(2):137-46. doi: 10.1007/s10840-011-9587-8. Epub 2011 May 26. PMID 21614530